CLINICAL TRIAL: NCT03935737
Title: Validation of a New Post Image Processing Engine (S-Vue™) for the Reduction of Ionizing Radiation Dose on X-ray Examination in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Susan D John, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-18-0348
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Chest X-ray for Clinical Evaluation
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Full dose Chest X-Ray: Subjects will receive a full (standard) dose chest X-ray at Day 1.
  Interventions: Diagnostic Test: Full Dose Chest X-Ray
- Low dose Chest X-Ray: Subjects will receive a follow up X-ray at at a lower dose within 3 months after the first dose.
  Interventions: Diagnostic Test: Low Dose Chest X-Ray

INTERVENTIONS:
Diagnostic Test: Full Dose Chest X-Ray — Full dose X ray at Day 1
  Other Names: GM85
  Groups: Full dose Chest X-Ray
Diagnostic Test: Low Dose Chest X-Ray — Low dose X ray within 3 months from full dose
  Other Names: GM85
  Groups: Low dose Chest X-Ray

SUMMARY:
The purpose of this study is to compare X-ray images obtained using the GM85 digital radiography machine at the standard full dose to X-ray images obtained using the GM85 digital radiography machine along with the Samsung S-Vue system, which is a image post-processing engine that allows images to be obtained using a lower dose. The study also aims to determine the lowest dose of radiation that can be used to get a good, readable x-ray of the chest in pediatric patients using Samsung S-Vue system.

ELIGIBILITY:
Inclusion Criteria:

* Standard weight/height outpatients who require two X-ray exams within 3 months in the US
* BMI is >5% and < 85% for participants over the age of 2;for participants less than 2 weight for length will be measured

Exclusion Criteria:

* Obese and underweight children as defined as BMI ,<5% or >85% according the World Health Organization growth chart for participants over 2 years of age; and for participants less than 2 years of age,weight for length will be measured

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients seen in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Image Quality as assessed by the Bureau of Radiological Health (BRH) method based scoring system-Anatomic landmark | baseline
  The BRH anatomic landmark score ranges from 0 to 100 with higher scores indicating better quality.
Image Quality as assessed by the Bureau of Radiological Health (BRH) method based scoring system-Anatomic landmark | within 3 months
  The BRH anatomic landmark score ranges from 0 to 100 with higher scores indicating better quality.
Image Quality as assessed by the Bureau of Radiological Health (BRH) method based scoring system-Physical parameters | baseline
  The BRH physical parameters score ranges from 0 to 100 with higher scores indicating better quality.
Image Quality as assessed by the Bureau of Radiological Health (BRH) method based scoring system-Physical parameters | within 3 months
  The BRH physical parameters score ranges from 0 to 100 with higher scores indicating better quality.

CONTACTS AND LOCATIONS:
Overall Officials: Susan D John, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No